CLINICAL TRIAL: NCT04883268
Title: Does Focusing on Body Functionality Improve Body Image Among Women Who Have Undergone Bariatric Surgery?
Brief Title: Focusing on Body Functionality After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Nederlandse Obesitas Kliniek (Unknown); Dutch Research Council (Unknown)
Responsible Party: Principal Investigator, Jessica Alleva, Assistant Professor, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ERCPN-167_03_05_2016
Record Dates: First submitted 2021-04-30; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Bariatric Surgery Candidate; Body Image

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants are randomised to group by the online research system. The investigator does not know what group participants have been assigned to. Participants are aware whether they have been assigned to the intervention or comparison (waitlist) group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group completed the Expand Your Horizon programme (Alleva et al., 2015).
  Interventions: Other: Expand Your Horizon
- Comparison Group (No Intervention): Participants in the comparison group did not complete any intervention (i.e., this was a waitlist comparison group).

INTERVENTIONS:
Other: Expand Your Horizon — Expand Your Horizon is an online programme, comprising three 15min writing exercises delivered over the course of 1 week. In each writing exercise, participants are asked to describe the functions of their body, and why those are personally meaningful to them.
  Arms: Intervention Group

SUMMARY:
This study investigated whether focusing on one's body functionality (i.e., everything the body can do, rather than how it looks) would lead to improvements in body image, self-esteem, and self-kindness among women who have undergone bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as female, being between 18 and 65 years old, having undergone bariatric surgery 5-7 months prior to the study, and qualifying for standard aftercare at the Nederlandse Obesitas Kliniek (NOK; Dutch Obesity Clinic).

Exclusion Criteria:

* N/A

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in appearance satisfaction over time (pretest, posttest, follow-ups) | Pretest (Day 1), posttest (Day 5), 1-week follow-up (Day 12), 3-month follow-up (Day 95)
  Appearance satisfaction was assessed using the Body Areas Satisfaction Subscale (BASS) of the Multidimensional Body-Self Relations Questionnaire (MBSRQ). Scores range from 1-5, with higher scores demonstrating higher appearance satisfaction.
Change in functionality satisfaction over time (pretest, posttest, follow-ups) | Pretest (Day 1), posttest (Day 5), 1-week follow-up (Day 12), 3-month follow-up (Day 95)
  Functionality satisfaction was assessed using the Physical Condition Subscale (PCS) of the Body Esteem Scale (BES). Scores range from 1-5, with higher scores demonstrating higher functionality satisfaction.
Change in body appreciation over time (pretest, posttest, follow-ups) | Pretest (Day 1), posttest (Day 5), 1-week follow-up (Day 12), 3-month follow-up (Day 95)
  Body appreciation was assessed using the Body Appreciation Scale-2 (BAS-2). Scores range from 1-5, with higher scores demonstrating higher body appreciation.
Change in body responsiveness over time (pretest, posttest, follow-ups) | Pretest (Day 1), posttest (Day 5), 1-week follow-up (Day 12), 3-month follow-up (Day 95)
  Body responsiveness was assessed using the Body Responsiveness Questionnaire (BRQ). Scores range from 1-7, with higher scores demonstrating higher body responsiveness.
Change in self-objectification over time (pretest, posttest, follow-ups) | Pretest (Day 1), posttest (Day 5), 1-week follow-up (Day 12), 3-month follow-up (Day 95)
  Self-objectification was assessed using the Self-Objectification Questionnaire (SOQ). Scores range from -25 to 25, with lower scores demonstrating higher levels of self-objectification.

SECONDARY OUTCOMES:
Changes in self-esteem over time (pretest, posttest, follow-ups) | Pretest (Day 1), posttest (Day 5), 1-week follow-up (Day 12), 3-month follow-up (Day 95)
  Self-esteem was assessed using the Rosenberg Self-Esteem Scale (RSE). Scores range from 10-40, with higher scores reflecting higher levels of self-esteem.
Changes in self-kindness over time (pretest, posttest, follow-ups) | Pretest (Day 1), posttest (Day 5), 1-week follow-up (Day 12), 3-month follow-up (Day 95)
  Self-kindness was assessed using the Self-Kindness Subscale (SKS) of the Self-Compassion Scale (SCS). Scores range from 1-7, with higher scores reflecting higher levels of self-kindness.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Alleva, Principal Investigator — Maastricht University; Carolien Martijn, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Maastricht University, Maastricht, Limburg
  - Nederlandse Obesitas Kliniek, Huis ter Heide, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Anonymised quantitative data (SPSS file) will be uploaded to DataVerse, and will be accessible upon request from the Principal Investigator. Study protocol and informed consent sheet will be available via ClinicalTrials.gov registration.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available as soon as the manuscript is published, with no deadline. The study protocol and informed consent sheet will be available immediately, with no deadline.
Access Criteria: Data will be available to other researchers for non-commercial purposes. Qualitative data (derived from participants' responses to the writing exercises) will not be shared, given the sensitive nature of the data, and given that participants did not provide consent for their writing exercises to be shared outside of the research team. Study protocol and informed consent sheet will be available for non-commercial purposes via ClinicalTrials.gov registration.
URL: https://dataverse.nl/

REFERENCES:
- [Background] Alleva JM, Martijn C, Van Breukelen GJ, Jansen A, Karos K. Expand Your Horizon: A programme that improves body image and reduces self-objectification by training women to focus on body functionality. Body Image. 2015 Sep;15:81-9. doi: 10.1016/j.bodyim.2015.07.001. Epub 2015 Aug 14. PMID 26280376
- [Derived] Alleva JM, Atkinson MJ, Vermeulen W, Monpellier VM, Martijn C. Beyond Body Size: Focusing on Body Functionality to Improve Body Image Among Women Who Have Undergone Bariatric Surgery. Behav Ther. 2023 Jan;54(1):14-28. doi: 10.1016/j.beth.2022.06.007. Epub 2022 Jul 3. PMID 36608971

DOCUMENTS (2):
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04883268/Prot_000.pdf
  • Informed Consent Form (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04883268/ICF_001.pdf